CLINICAL TRIAL: NCT01639391
Title: Creation of a Bank of Fibroblast From Patients With Amyotrophic Lateral Sclerosis: Pilot Study
Acronym: ALSCELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2010-33
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients (Experimental)
  Interventions: Procedure: skin biopsy

INTERVENTIONS:
Procedure: skin biopsy — biopsy 5mm maximum on healthy skin under local anaesthesia.

SUMMARY:
Patients with ALS will be included in the reference center for ALS in hospital La Pitié Salpêtrière, Paris.

The study proposes to investigate the pathophysiology of ALS by setting up a fibroblast bank for studying molecular, cellular and genetic parameters of the pathology.

iPS (induced pluripotent stem cells) and then differentiated cells will be generated.

The pathophysiology of ALS will be studied on the 3 types of cells (fibroblasts, iPS, differentiated cells).

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* ALS sporadic or familial or unknown

Exclusion Criteria:

* known cutaneous disease not allowing the biopsy
* platelets less than 10 000/m3
* suspected or known xylocain allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-11-29 (Actual); Primary Completion 2015-03-17 (Actual); Study Completion 2015-03-17 (Actual)

PRIMARY OUTCOMES:
Success of fibroblast culture, amplification, and freezing pellets | 2 months

SECONDARY OUTCOMES:
Induced pluripotent Stem Cells generation success | 2 years
neurones, motoneurones, glial cells obtention from fibroblasts or iPS | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lucette Lacomblez, MD, Principal Investigator — hôpital La Pitié Salpêtrière, Paris; Delphine Bohl, PhD, Study Chair — Institut Pasteur
Locations (1):
- Centre référent maladies rares SLA, Paris, France